CLINICAL TRIAL: NCT03166462
Title: Effects of Obstructive Sleep Apnea in Elective Orthopaedic Surgery
Brief Title: Obstructive Sleep Apnea in Elective Orthopaedic Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding and clinical resources
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Victor Hugo Hernandez, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20160732
Record Dates: First submitted 2016-09-07; First posted 2017-05-25 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Sleep Apnea, Obstructive; Total Knee Arthroplasty; Total Hip Arthroplasty
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in this arm will proceed through the current standard of care for pre-operative screening performed by either the patient's primary care physician or the "pre-operative" anesthesia clinic which screens patients prior to total knee or total hip arthroplasty.
- Intervention (Experimental): Patients in this arm will be referred to the Sleep Medicine clinic at the University of Miami Hospital for additional testing and evaluation for obstructive sleep apnea. If they are successfully diagnosed, they will receive appropriate treatment and any interventions for the peri-operative period as recommended by the pulmonary medicine team.
  Interventions: Other: Evaluation by Sleep Medicine Specialists

INTERVENTIONS:
Other: Evaluation by Sleep Medicine Specialists — Patients randomized to the intervention arm will be referred to the sleep medicine specialists for evaluation. All of their recommendations will be followed if indicated.
  Arms: Intervention

SUMMARY:
Demand for Total Knee Arthroplasty (TKA) and Total Hip Arthroplasty (THA) is increasing steadily and is projected to continue trending upwards in the coming years. Concomitant with that trend is the increase in prevalence of obesity. Obesity serves as a common risk factor for osteoarthritis, obstructive sleep apnea and medical complications.

Obstructive Sleep Apnea (OSA) is defined as episodes of obstructive apneas and hypopneas during sleep, with daytime somnolence. It occurs commonly in obese, middle age and elderly men and has an estimated prevalence of 5% - 9%.

Pre-operative screening for elective surgical procedures is a critical component of a successful surgical outcome. Patients with medical comorbidities ideally will undergo medical treatment or optimization to minimize the risk peri-operatively and post-operatively. Obstructive sleep apnea has been shown in numerous studies to be a risk factor for cardiopulmonary complications following surgery. The contributing factors include alterations in REM sleep post-operatively and opioid induced respiratory suppression post-operatively.

The STOP-BANG patient questionnaire is a validated patient survey that uses both objective and subjective data to screen patients for their risk of OSA. The sensitivity of the STOP-BANG questionnaire for moderate-to-severe OSA has been estimated as high as 97.74%. Authors have also shown that higher STOP-BANG scores are independently associated with increased risk for post-operative complication.

Other authors have utilized similar pre-operative questionnaires to screen for occult pulmonary disease in patients scheduled for elective joint arthroplasty. They found a slightly increased incidence of OSA in this population as compared with the national average, over 50% of which were previously undiagnosed.

The American Society of Anesthesiologists task force on perioperative management of patients with OSA published extensive guidelines aimed at reducing morbidity and mortality. Improved diagnosis pre-operatively could aid in proper compliance with these guidelines. These recommendations include preferential use of regional analgesia, reduction in systemic opioids, monitoring of oxygen saturation and nonsupine posture.

The mainstay of treatment for OSA is a positive pressure airway device such as Continuous Positive Airway Pressure (CPAP) or in severe cases Nasal Intermittent Positive Pressure Ventilation (NIPPV). Post-operatively continuation of these treatments in patients with known OSA is often recommended. Some authors have demonstrated reductions in Apnea-Hypopnea Index postoperatively through the use of CPAP.

However, a recent meta-analysis evaluating the effect of pre-operative or post-operative CPAP in patients with OSA concluded that the use of CPAP did not reduce post-operative adverse events.

Given the projected increase in demand for joint arthroplasty, the ever-increasing incidence of obesity, the ambiguity surrounding the topic and the potential to clinically impact post-operative morbidity, mortality and health care costs, shows the need for further studies.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Have signed the written informed consent form
* STOP-BANG score greater than or equal to 5

Exclusion Criteria:

* Patients not fluent in the language of the informed consent form (English, Spanish, Creole)
* Prisoners
* Pregnancy
* Reported to have mental illness or belonging to a vulnerable population
* Patients with previous diagnosis and treatment of Obstructive sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-02-08 (Estimated); Study Completion 2018-02-08 (Estimated)

PRIMARY OUTCOMES:
Post Operative Complications both acute and short term | 90 days
  The investigators will assess if screening and subsequent treatment for obstructive sleep apnea reduces the incidence of unplanned admission to the intensive care unit, post operative delirium, post operative hypoxia necessitating supplemental oxygen, myocardial infarction as measured by objective measures such as troponin levels and EKG changes and thromboembolism. The incidence of any one of these factors is relatively low. Therefore the investigators will aggregate them as the number of subjects needed to asses them individually would be too large.

SECONDARY OUTCOMES:
Financial Impact | 90 days
  Readmission Rate
Financial Impact | 30 days
  Length of inpatient stay postoperatively
Financial Impact | 90 days
  Discharge location: Home versus skilled nursing facility versus inpatient rehabilitation versus long term care facility versus other
Functional Outcomes | 90 days
  Oxford Hip/Knee Score measured in units of the scale
Functional Outcomes | 90 days
  Western Ontario and McMaster Universities Arthritis Index measured in units of the scale, WOMAC
Functional Outcomes | 90 days
  Harris Hip/Knee Score measured in units of the scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided